CLINICAL TRIAL: NCT00919347
Title: The Relative Prevalence and Severity of Autonomic Nervous System Dysfunction in Diabetic Patients Undergoing Retinal Surgery
Brief Title: The Relative Prevalence and Severity of Autonomic Nervous System Dysfunction
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gwendolyn L. Boyd, MD, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F080909006
Record Dates: First submitted 2009-06-01; First posted 2009-06-12 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Cardiovascular Autonomic Neuropathy; Diabetic Autonomic Neuropathy; Autonomic Dysfunction
Keywords: Cardiovascular Autonomic Neuropathy; Diabetic Autonomic Neuropathy; Autonomic Dysfunction
MeSH Terms: conditions — Diabetic Neuropathies; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: ANSAR ANX 3.0 Software — Three values are calculated by the ANSAR ANX 3.0® software of the spectral analysis of HRV and respiration:
  1. RFa an indicator of parasympathetic function with normal values between 0.5 and 10 bpm2;
  2. LFa an indicator of sympathetic function also with normal values between 0.5 and 10 bpm2;
  3. SB or the ratio of LFa/RFa with normal reference values of 0.4 to 3.0.
  The ANSAR ANX 3.0® software defines three different levels of autonomic neuropathy (autonomic dysfunction) as follows (see Figure 1):
  * Cardiovascular Autonomic Neuropathy (CAN): resting parasympathetic insufficiency (not enough parasympathetic protection for the heart) or RFa < 0.1 bpm2.
  * Diabetic Autonomic Neuropathy (DAN), or advanced autonomic dysfunction in non-diabetics, is defined as low autonomics: LFa < 0.5 bpm2 or 0.1 < RFa < 0.5 bpm2.
  * Autonomic Dysfunction: normal resting LFa and RFa, but low LFa response to Valsalva or low RFa response to deep breathing.

SUMMARY:
The purpose of this study is to measure the prevalence and severity of cardiac autonomic neuropathy (CAN), diabetic autonomic neuropathy (DAN) which in non-diabetics is termed advanced nervous system (ANS) dysfunction, and autonomic dysfunction as well as the overall sympathovagal balance (SB) in the CEFH population of diabetic patients versus non-diabetic patients undergoing elective vitreoretinal surgery.

DETAILED DESCRIPTION:
The purpose of this study is to measure the prevalence and severity of cardiac autonomic neuropathy (CAN), diabetic autonomic neuropathy (DAN) which in non-diabetics is termed advanced nervous system (ANS) dysfunction, and autonomic dysfunction as well as the overall sympathovagal balance (SB) in the CEFH population of diabetic patients versus non-diabetic patients undergoing elective vitreoretinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Type I and Type II Diabetic patients 19 or older who are scheduled for elective surgery to improve vision impaired by diabetic retinopathy
* Patients scheduled during the same time period without diabetes for retinal surgery will serve as an age and gender matched reference group to undergo the non-invasive ANS testing on the day of surgery

Exclusion Criteria:

* Inability to stand will only do baseline, deep breathing and Valsalva portions (A-D) of the testing as described in section 8.1
* Patients with syncope on standing will only do portions A-D of the test
* Inability to cooperate with deep breathing and Valsalva
* Tracheoscopy or otherwise not able to perform a Valsalva
* Not desiring to participate after informed consent
* Known history of idiopathic dysautonomia
* Pulmonary difficulties associated with hyperventilation, including acute URI
* Pacemaker dependent
* Persistently high intraocular pressure despite treatment
* Atrial fibrillation
* Ventricular arrhythmias greater than 10 beats per minute
* Taking MAO inhibitors

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patiented from the Callahan Eye Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be to quantify, using the ANSR ANX 3.0 technology, the prevalence of cardiac autonomic neuropathy (CAN), diabetic autonomic neuropathy (DAN),referred to as advanced autonomic nervous system dysfunction in non-diabetic patients. | 15 minutes

SECONDARY OUTCOMES:
The strength of various comorbidities as predictors of autonomic dysfunction in both diabetics and non-diabetics will be evaluated. The differential effect of these various comorbidities in Type I versus Type II diabetes on ANS dysfunction and neuropathy | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Callahan Eye Foundation Hospital, Birmingham, Alabama, United States